CLINICAL TRIAL: NCT02799043
Title: Randomized Evaluation of Redo Ablation Procedures of Atrial Fibrillation With Focal Impulse and Rotor Modulation Guided Procedures (REDO-FIRM)
Brief Title: Randomized Evaluation of Redo Ablation Procedures of Atrial Fibrillation With FIRM Guided Procedures
Acronym: REDO-FIRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: REDO-FIRM
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Persistent Atrial Fibrillation; Paroxysmal Atrial Fibrillation
Keywords: FIRMap, Rotor, FIRM-guided procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard PVI (Active Comparator): Standard catheter ablation including pulmonary vein isolation (PVI) procedure.
  Interventions: Procedure: Standard PVI
- FIRM-guided Procedure and PVI (Experimental): FIRM-guided procedure followed by PVI.
  Interventions: Procedure: FIRM-Guided Procedure and PVI

INTERVENTIONS:
Procedure: Standard PVI — Standard PVI procedure without FIRMap.
  Other Names: Pulmonary vein isolation; Ablation; Arrhythmia; Atrial fibrillation Mapping
  Arms: Standard PVI
Procedure: FIRM-Guided Procedure and PVI
  Other Names: Pulmonary vein isolation; Atrial fibrillation Mapping; FIRMap
  Arms: FIRM-guided Procedure and PVI

SUMMARY:
A prospective, multicenter, randomized study to assess the safety and effectiveness of FIRM-guided procedures in conventional "redo" RF ablation procedures for the treatment of persistent and paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The hypothesis of this study was that Focal Impulse and Rotor Modulation (FIRM) guided procedures will eliminate the source of clinical arrhythmias in subjects with clinical indications for repeat AF ablation procedures.

This study is a prospective, multicenter, randomized, controlled study to assess the safety and effectiveness of FIRM procedures followed by ablation including pulmonary vein isolation versus a standard conventional procedure including pulmonary vein isolation for the redo-treatment of persistent or paroxysmal atrial fibrillation after one failed previous pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing at least one (1) documented episode of spontaneous persistent or paroxysmal atrial fibrillation during the last 3 months by rhythm strip/ECG.
* One (1) previous AF ablation (PVI-only - any technology) after Jan-01-2013, but NOT within the last 3 months.
* Left atrial diameter < 6.0 cm via transthoracic echo or transesophageal echo; or <6.5 cm via CT or MRI with 6 months prior to the procedure.
* Sustained spontaneous or induced AF (>5 min uninterrupted).

Exclusion Criteria:

* Presence of structural heart disease with clinical significance
* NYHA Class IV
* Ejection fraction < 35%
* Previous AF ablation within the last 3 months
* ASD closure device, LAA closure device, prosthetic mitral or tricuspid valve, or permanent pacemaker.
* History of myocardial infarction (MI) within the past three (3) months
* Atrial clot/thrombus noted within 72 hours of the procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Stefan G. Spitzer, MD, Principal Investigator — Praxisklinik Herz und Gefäße Dresden, Germany
Locations (24):
- United States (12):
  - Arizona Heart Rhythm Research Cente, Phoenix, Arizona
  - Ventura Cardiology Consultants, Ventura, California
  - Broward Health, Fort Lauderdale, Florida
  - St. Vincent's HealthCare, Jacksonville, Florida
  - Loyola University, Chicago, Illinois
  - Northwestern University - Bluhm Cardiovascular Institute, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Heart, Falls Church, Virginia
- University Hospital of Antwerp, Antwerp, Flanders, Belgium
- Germany (10):
  - Klinikum Coburg, Coburg, Bavaria
  - Furth Medical Clinic for Heart and Lung Diseases, Fürth, Bavaria
  - The Dr. Müller Kliniken, Munich, Bavaria
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam, Brandenburg
  - Kardiocentrum Frankfurt, Frankfurt, Main
  - Leipzig Heart Institute GmbH, Leipzig, Saxony
  - Luebeck University Heart Center, Lübeck, Schleswig-Holstein
  - Ruhr University Bochum - Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen
  - UKB (Unfallkrankenhaus Berlin), Berlin
  - Praxisklinik Herz und Gefäße Dresden, Dresden
- Medical Center Rotterdam (Erasmus MC), Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In order to be randomized, subjects must have met the following criteria:
  1. Atrial Fibrillation is sustained for at least 5 minutes uninterrupted.
  2. Confirmation of Pulmonary Vein reconnection. If Atrial Fibrillation could not be sustained or if Pulmonary Vein reconnection could not be confirmed, the patient was disqualified and were not randomized / enrolled in the study.
Groups:
- FIRM-guided Procedure and PVI: FIRM-guided procedure followed by PVI.
  FIRM-Guided Procedure and PVI
Period: Overall Study
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI
Started | 133 | 136
Treated (Intention to treat population.) | 131 | 134
Completed | 122 | 121
Not Completed | 11 | 15
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Moved to different country | 0 | 1
Not completed — Trial Screen Failure | 1 | 0
Not completed — Failed Inclusion/Exclusion Criteria | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI | Total
Number analyzed (Participants) | 133 | 136 | 269
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.0 [58 to 70] | 65.5 [59 to 70] | 65 [59 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 37 | 92
  Male | 78 | 99 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 131 | 135 | 266
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 0 | 0 | 0
  White | 131 | 133 | 264
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Netherlands | 13 | 11 | 24
  Belgium | 2 | 4 | 6
  United States | 20 | 27 | 47
  Germany | 98 | 94 | 192

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Atrial Fibrillation Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atrial Flutter (AFL) Recurrence at 12 Months Post Procedure.
Description: Single procedure freedom from recurrence from 3-12 months post procedure
Time Frame: 12 months post procedure
Population: Intention to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 122 | 120
Participants | 72 | 76

2. Primary Outcome: Freedom From Serious Adverse Events Related to the Procedure
Description: Freedom from any procedure-related serious adverse event from 0-10 days post procedure
Time Frame: 10-day post procedure
Population: Intention to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 128 | 134
Participants | 120 | 125

3. Primary Outcome: Freedom From Serious Adverse Events Related to the Procedure
Description: Freedom from any procedure-related serious adverse event from 0-12 months post procedure
Time Frame: 12-month post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI
Number analyzed (Participants) | 121 | 121
Participants | 113 | 107

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard PVI | FIRM-guided Procedure and PVI
All-Cause Mortality (participants affected / at risk) | 1/131 | 2/134
Serious Adverse Events (participants affected / at risk) | 8/131 | 14/134
Other Adverse Events (participants affected / at risk) | 0/131 | 0/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard PVI (N=131) | FIRM-guided Procedure and PVI (N=134)
Vascular pseudoaneurysm (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Anesthetic complication (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Catheter site hemorrhage (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral infarction (Vascular disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Dyspnea (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Esophageal stent insertion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Peripheral artery stenosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Prostatitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT02799043/Prot_SAP_000.pdf